CLINICAL TRIAL: NCT01131884
Title: Double Blind Placebo Controlled Trial to Evaluate Preservation of Bone Mineral Density of the Hip and Distal Femur by Biphosphate Therapy (Fosamax) Following Spinal Cord Injury
Brief Title: Pilot Study of Fosamax in Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Only 1 participant enrolled since the beginning of this study
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, K. R Poduri, Chair of Department of PM&R, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U of R 29563
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Spinal Cord Injury; Osteoporosis
Keywords: ASIA A or ASIA B Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries; Osteoporosis | interventions — Alendronate; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fosamax (Active Comparator): Fosamax at 70 mgs q weekly by mouth for the duration of the study.
  Interventions: Drug: Fosamax
- Placebo Sugar Pill (Placebo Comparator): Double blind study using Fosamax versus placebo. Placebo is an inactive drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fosamax — 70mg of Bisphosphonate therapy (Fosamax) will be taken weekly for a year
  Other Names: Alendronate sodiuum
  Arms: Fosamax
Drug: Placebo — Placebo is an inactive pill that will look similar to the active drug. You will not know whether you are receiving active drug or placebo.
  Other Names: Sugar pill
  Arms: Placebo Sugar Pill

SUMMARY:
Study is designed to evaluate the efficacy of oral fosamax in prevention on osteoporosis in acute spinal cord injury. Efficacy will be measured by a duel energy X-Ray absorptiometry (DEXA) scan every 6 months. Patients will complete 3 visits, screening, 6 months, 12 months and be required to take oral fosamax versus placebo weekly.

DETAILED DESCRIPTION:
The project was funded on August 13, 2009 and was awarded to one of our trainees, Dr. Matthew Abraham, a PGY3 in our program and our IRB approval was obtained with much time and effort on February 24, 2010. We followed the protocol and so far we recruited just one patient on September 19, 2011 who completed the study but we encountered with many unexpected obstacles to recruit any more patients to the study. The main obstacle was that the spine surgeons' refusal to start the study drug for months after surgery for fear of complications with wound healing. Secondly, the few appropriate and eligible patients we tried to recruit declined to participate.

We were unable to recruit any more patients to this study and hence the study was closed.

The one patient that was recruited completed the study. Since it is only one subject in the study, no conclusions can be drawn.

ELIGIBILITY:
Inclusion Criteria:

* American Spinal Cord Injury Association (ASIA) A or American Spinal Cord Injury Association (ASIA) B Spinal Cord Injury

Exclusion Criteria:

* History of hypersensitivity to alendronate or other bisphosphonates
* esophageal abnormality
* inability to sit/stand upright for 30 minutes
* creatinine clearance less than 35 milliliters/minute
* hypothyroidism
* malignancy
* pregnancy
* prolonged steroid use

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanakadurga R Poduri, M.D., Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - University of Rochester Physical Medicine and Rehabilitation, Rochester, New York
  - University of Rochester, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A 57 year old T4 paraplegic was recruited while he was going through rehabilitation at Strong Memorial Hospital inpatient rehab unit. This patient was recruited and signed consent on 8/05/2011.He underwent lab work and dexa scan per protocol and on completion of the investigation on September 19, 2011 he started the treatment(Fosamax vs. Placebo).
Pre-assignment Details: Recruitment beyond one patient was not possible due to A. surgeons unwillingness to initiate Fosomax treatment for fear of wound healing. B. The eligible patients' reluctance to participate in the study. C. Given the length of time it took to enroll one, it is not feasible to complete the study with required # in the protocol in the next few years
Groups:
- Fosamax: Fosamax : 70mg of Bisphosphonate therapy (Fosamax) will be taken weekly for a year
- Placebo Sugar Pill: Double blind study using Fosamax versus placebo. Placebo is an inactive drug.
  Placebo : Placebo is an inactive pill that will look similar to the active drug. You will not know whether you are receiving active drug or placebo.
Period: Overall Study
Arm/Group | Fosamax | Placebo Sugar Pill
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosamax | Placebo Sugar Pill | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (0) |  | 58 (0)
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density
Description: Whether or not Fosamax increases bone mineral density at the hip and distal femur in spinal cord injury induced osteoporosis
Time Frame: 1 year after enrollment
Population: No analysis performed as there was only one patient who participated in this study
Arm/Group | Fosamax | Placebo Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Fosamax | Placebo Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No